CLINICAL TRIAL: NCT04439279
Title: MATCH Treatment Subprotocol R: Phase II Study of Trametinib in Patients With BRAF Fusions, or With NonV600E, Non-V600K BRAF Mutations
Brief Title: Testing Trametinib as a Potential Targeted Treatment in Cancers With BRAF Genetic Changes (MATCH-Subprotocol R)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03272; NCI-2020-03272 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-R (Other: ECOG-ACRIN Cancer Research Group); EAY131-R (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (trametinib) (Experimental): Patients receive trametinib dimethyl sulfoxide PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Trametinib Dimethyl Sulfoxide

INTERVENTIONS:
Drug: Trametinib Dimethyl Sulfoxide — Given PO
  Other Names: Mekinist; Meqsel; Spexotras

SUMMARY:
This phase II MATCH treatment trial identifies the effects of trametinib in patients with cancer having genetic changes called BRAF mutations and fusions. Trametinib may block proteins called MEK1 and MEK2, which may be needed for growth of cancer cells that express BRAF mutations. Researchers hope to learn if giving trametinib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive trametinib dimethyl sulfoxide (trametinib) orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have a BRAF non-V600 mutation or BRAF fusion, or another aberration, as identified via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have NONE of the following cardiac criteria:

  * Clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
* Patients must have an echocardiogram (ECHO) or a nuclear study (multigated acquisition scan [MUGA] or First Pass) within 4 weeks prior to registration to treatment and must not have a left ventricular ejection fraction (LVEF) < the institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible
* Patients who previously received monoclonal antibody therapy (e.g. ipilimumab, nivolumab, pembrolizumab and others) must have stopped the prior therapy for 8 or more weeks before starting on trametinib

Exclusion Criteria:

* Patients with a history of interstitial lung disease or pneumonitis are excluded
* Patients must not have known hypersensitivity to trametinib or compounds of similar chemical or biologic composition or to dimethyl sulfoxide (DMSO)
* Patients must not have a history or current evidence/risk of retinal vein occlusion (RVO). An eye exam is required at baseline
* Patients who previously received MEK inhibitors (including, but not limited to, trametinib, binimetinib, cobimetinib, selumetinib, RO4987655 (CH4987655), GDC-0623 and pimasertib) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B Johnson, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol R was activated on August 12, 2015. A total of 50 patients were assigned to this arm after screening, 48 from screening cohort and 2 from outside assay. Of the 50 patients, 35 patients were enrolled to arm R between December 4, 2015 and August 17, 2017.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For the subprotocol R, patients had to have BRAF fusion or Non-V600E, Non-V600K mutations.
Groups:
- Subprotocol R: Patients receive trametinib dimethyl sulfoxide PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Subprotocol R
Started | 35
Started Protocol Therapy | 35
Eligible | 33
Reported Adverse Events Data | 34 (Adverse event was not assessed on one patient before discontinuing therapy due to withdraw/refusal)
Completed | 0 (Treatment continued until disease progression or intolerability.)
Not Completed | 35
Not completed — Adverse Event | 7
Not completed — Death | 4
Not completed — Disease progression | 17
Not completed — Complicating disease | 3
Not completed — Withdrawal by Subject | 2
Not completed — Ineligible | 1
Not completed — Treatment still ongoing | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Subprotocol R
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 65 [40 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) among all eligible and treated patients. Best overall response was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. The 90% two-sided binomial exact confidence interval was calculated for ORR.
Time Frame: assessed at baseline, then every 2 cycles until disease progression, up to 3 years post registration
Population: eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Subprotocol R
Number analyzed (Participants) | 33
percentage of participants | 3 [0.1 to 16]

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. The 6-month PFS rate was estimated using the Kaplan-Meier method which can provide a point estimate for any specific time point. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients.
Time Frame: assessed at baseline, then every 2 cycles until disease progression, up to 3 years post registration
Population: eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Subprotocol R
Number analyzed (Participants) | 33
percentage of participants | 20 [10 to 33]

3. Secondary Outcome: Progression-free Survival
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients.
Time Frame: assessed at baseline, then every 2 cycles until disease progression, up to 3 years post registration
Population: eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Subprotocol R
Number analyzed (Participants) | 33
months | 1.8 [1.6 to 3.4]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years
Description: All 35 patients enrolled to the trial were monitored for mortality, 34 patients were monitored for adverse events as one patient refused to submit adverse event data right after starting the protocol therapy.
Arm/Group | Subprotocol R
All-Cause Mortality (participants affected / at risk) | 9/35
Serious Adverse Events (participants affected / at risk) | 14/34
Other Adverse Events (participants affected / at risk) | 29/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subprotocol R (N=34)
Anemia (Blood and lymphatic system disorders) | 5
Sudden death NOS (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Ejection fraction decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subprotocol R (N=34)
Anemia (Blood and lymphatic system disorders) | 10
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2
Chills (General disorders) | 2
Edema limbs (General disorders) | 12
Fatigue (General disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 5
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 7
Paronychia (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 10
Ejection fraction decreased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 4
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Dizziness (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT04439279/Prot_000.pdf